CLINICAL TRIAL: NCT02165852
Title: A Prospective Comparative Study of Papillectomy
Brief Title: Comparison on the Efficacy of Endoscopic Snare Papillectomy With or Without Submucosal Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Soon Chun Hyang University (Other)
Responsible Party: Principal Investigator, Tae Hoon Lee, MD, Soon Chun Hyang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Papillectomy Study
Record Dates: First submitted 2014-03-25; First posted 2014-06-18 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Ampulla of Vater Adenoma
Keywords: ampulla of Vater; adenoma; papillectomy; injection; non-injection
MeSH Terms: conditions — Adenoma | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Papillectomy without injection (Experimental): Conventional snaring mucoal resection without submucosal injection
  Interventions: Procedure: Papillectomy without injection
- Papillectomy with injection (Active Comparator): Conventional mucosal resction method following injeciton of diluted epinephrine mixture.
  Interventions: Procedure: Papillectomy with injection

INTERVENTIONS:
Procedure: Papillectomy without injection — Conventional endoscopic mucosal resection of ampulla of Vater using a snare with electrocurrent.
  Arms: Papillectomy without injection
Procedure: Papillectomy with injection — Conventional endoscopic mucosal resection of ampulla of Vater without submucosal saline or diluted epinephrine injection.
  Arms: Papillectomy with injection

SUMMARY:
Because the ampulla of Vater is strategically located at the confluence of the pancreatic and common bile ducts, endoscopic resection of papillary neoplasms may be technically different from endoscopic mucosal resection in other parts of the gastrointestinal tract. The best method of endoscopic ablation and the optimal period for surveillance have not been established.

DETAILED DESCRIPTION:
While some endoscopists advocate the use of submucosal injection of either physiologic saline solution or dilute epinephrine, some do not. Whether physiologic saline solution or dilute epinephrine should be used is also not established. Submucosal injection of either dilute epinephrine or saline solution may be useful for avoiding inappropriate resection because failure to lift the tumor from the proper muscle layer of the duodenum may indicate deeper invasion18 and is the strongest predictor of malignancy.

In adenomas of the major duodenal papilla, however, some investigators do not recommend submucosal injection. Not only the surrounding mucosa at the region of the duodenal papilla but also the tumor is lifted by submucosal injection, so capturing the lesion with a snare becomes difficult.

ELIGIBILITY:
Inclusion Criteria:

* ampulla of Vater adenoma
* no uncontrolled coagulopathy

Exclusion Criteria:

* adenocarcinoma of ampulla of Vater
* uncontrolled coagulopathy
* refusal to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
complete resection | one month
  Following endoscopic papillectomy, complete resection will be estimated by pathologic examination

SECONDARY OUTCOMES:
complication | within 24 hours
  Immediate complications after papillecotmy Delayed complications during 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tae Hoon Lee, MD, PhD, Principal Investigator — SoonChunHyang University School of Medicine
Locations (1):
- Soonchunhyang University Cheonan Hospital, Cheonan, South Korea

REFERENCES:
- [Derived] Hyun JJ, Lee TH, Park JS, Han JH, Jeong S, Park SM, Lee HS, Moon JH, Park SH. A prospective multicenter study of submucosal injection to improve endoscopic snare papillectomy for ampullary adenoma. Gastrointest Endosc. 2017 Apr;85(4):746-755. doi: 10.1016/j.gie.2016.08.013. Epub 2016 Aug 24. PMID 27566056